CLINICAL TRIAL: NCT05242380
Title: The Effects of Kettlebell Exercise Training in Patients With Pulmonary Arterial Hypertension
Brief Title: Exercise Training in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Pinar BASTURK, Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-152558
Record Dates: First submitted 2021-12-25; First posted 2022-02-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kettlebell Exercise (Experimental): 8-week, 3-day/week supervised training will be applied to the participants in this group. After the initial assessment, patients in this group will receive a one-session education on the pathophysiology of PAH, the benefits of physical activity, and energy conservation techniques during activities of daily living. Pharmacological treatment of patients in this group will be continued.
  Interventions: Other: Kettlebell Exercise
- Control (No Intervention): Any intervention will not be performed. After the initial assessment, patients in this group will receive a one-session education on the pathophysiology of PAH, the benefits of physical activity, and energy conservation techniques during activities of daily living. Pharmacological treatment of patients in this group will be continued.

INTERVENTIONS:
Other: Kettlebell Exercise — The exercise training plan for this group consists of 4 stages. Each stage lasts 2 weeks and consist of 5 kettlebell (KB) exercises. These exercises will continue from basic (single movement training) to advanced (comprehensive movement training) and is geared towards functional training. Participants will perform 2 sets of 12 repetitions of each exercise. Each training session is planned to last 45 minutes.
  The following exercises will be used in KB training: biceps curl, triceps extension, kettlebell swing (two-handed), kettlebell dead lift, kettlebell goblet squat, suitcase carry, waiter carry, bottoms up carry, farmer's walk, overhead carry, lunge, kettlebell row.
  Arms: Kettlebell Exercise

SUMMARY:
In this study, the effects of kettlebell exercise training on functional capacity, dyspnea and activities of daily living in patients diagnosed with Pulmonary Arterial Hypertension (PAH) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pulmonary arterial hypertension (PAH) by a specialist physician in accordance with the 2015 guideline for the treatment and diagnosis of pulmonary hypertension of the European Heart and Respiratory Societies (ERS/ESC),
* Patients with stable pharmacological treatment,
* Patients clinically stable at least last three months.

Exclusion Criteria:

* Presence of orthopedic or neurological problems that will affect functional tests and muscle strength measurement,
* Recent surgical procedures,
* Recent syncope,
* Pregnancy,
* Presence of severe left heart failure,
* Presence of severe ischemic heart disease,
* Hypertensive patients,
* Patients who have problems in communicating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Task related oxygen uptake | 8 weeks
  Cardiopulmonary data will be evaluated with mobile cardiopulmonary exercise test during daily activities. Participants will perform the following activities with mobile cardiopulmonary exercise test (CPET): putting on socks on both feet (sitting on a chair), putting on both shoes (sitting on a chair), putting on a coat (while standing), lifting material (placing 6 jars -each 400 gram- at chest-level height), sweeping the floor for 4 minutes, washing dishes for 4 minutes, go up and down stairs - 1 floor. There will be a 5 minute rest between all activities.
Functional capacity | 8 weeks
  The 6-minute walk test will be performed.
Peripheral muscle strength | 8 weeks
  Isometric muscle strength will be measured with a handheld dynamometer for elbow flexion, knee extension, knee flexion, shoulder flexion, shoulder abduction, hip flexion and m.serratus anterior.
Handgrip strength | 8 weeks
  Hand grip strength will be measured with a digital hand dynamometer.

SECONDARY OUTCOMES:
Activity status | 8 weeks
  This outcome will be assessed with the Duke Activity Status Index. As a result of scoring, a total score ranging from 0 to 58.2 is obtained. Higher scores indicate higher functional capacity.
Health-related quality of life | 8 weeks
  This outcome will be assessed with the emPHasis-10. emPHasis-10 consists of 10 items and results in a score out of 50, where a higher score represents a higher symptom burden.
Activities of daily living | 8 weeks
  This outcome will be assessed with the London Chest Activity of Daily Living Scale. It is a questionnaire consisting of fifteen items. Each item is given a score ranging from 0 to 5. Higher scores indicate greater limitation in activities of daily living. The total score can reach a maximum of 75
Sleep quality | 8 weeks
  This outcome will be assessed with the Pittsburgh Sleep Quality Index. The questionnaire consists of 19 individual items. Each item is given a score ranging from 0 to 3, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, PhD, PT, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Institute of Cardiology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen HT, Wu HJ, Chen YJ, Ho SY, Chung YC. Effects of 8-week kettlebell training on body composition, muscle strength, pulmonary function, and chronic low-grade inflammation in elderly women with sarcopenia. Exp Gerontol. 2018 Oct 2;112:112-118. doi: 10.1016/j.exger.2018.09.015. Epub 2018 Sep 20. PMID 30243898
- [Background] Spruit MA, Wouters EF, Eterman RM, Meijer K, Wagers SS, Stakenborg KH, Uszko-Lencer NH. Task-related oxygen uptake and symptoms during activities of daily life in CHF patients and healthy subjects. Eur J Appl Physiol. 2011 Aug;111(8):1679-86. doi: 10.1007/s00421-010-1794-y. Epub 2011 Jan 6. PMID 21210281
- [Background] Mapelli M, Salvioni E, Bonomi A, Gugliandolo P, De Martino F, Vignati C, Berna G, Agostoni P. How Patients With Heart Failure Perform Daily Life Activities: An Innate Energy-Saving Strategy. Circ Heart Fail. 2020 Nov;13(11):e007503. doi: 10.1161/CIRCHEARTFAILURE.120.007503. Epub 2020 Nov 17. PMID 33201750
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941